CLINICAL TRIAL: NCT00774722
Title: Phase 2 Study Evaluation of Topical 10% Metronidazole Ointment for the Reduction of Pain After Haemorrhoidectomy
Brief Title: A Randomised Controlled Trial of the Use of Topical Metronidazole (10%) to Reduce Pain After Haemorrhoidectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: S.L.A. Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MET/02; EudraCT Number 2005-001396-35
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Haemorrhoidectomy
MeSH Terms: interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metronidazole (Experimental)
  Interventions: Drug: Metronidazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — 10% ointment, three times daily for 14 days

SUMMARY:
The purpose of this study is to determine whether metronidazole 10% ointment , applied topically three times a day in and around the anus, on the reduction of pain following haemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Have Grade 3 or 4 haemorrhoids (external disease with or without significant internal component)
* Be scheduled for diathermy haemorroidectomy with ≥2 quadrant involvement
* Be medically fit for surgery
* Subjects must be aged 18 years or over and of the legal age of consent.
* If female, the subject must not be lactating and must be (a) post-menopausal, (b) surgically sterilised, or (c) have a negative pregnancy test result prior to entry into the study and will use adequate contraception for the duration of the study.
* Must have provided written informed consent to participate.

Exclusion Criteria:

* They have had surgery to the anus or rectum in the past 8 weeks
* Suffer from a chronic pain syndrome which requires regular narcotic analgesia
* Have anal fissures
* Have diagnosed Crohn's disease
* Allergic to metronidazole
* Are taking any prohibited medication.
* Deemed mentally incompetent
* Considered by their physician unlikely to be able to comply with the protocol.
* Taken part in an experimental drug study in the preceding three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the efficacy of 10% metronidazole ointment in reducing post-operative pain associated with haemorrhoidectomy as compared to placebo. | 14 days

SECONDARY OUTCOMES:
evaluate and compare the expected pain following haemorrhoidectomy in the treatment and placebo groups. overall patient satisfaction with the operation. the number of analgesics required post-operatively the time taken to return to work and/or | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Jordan, BSc, Study Director — SLA Pharma
Locations (5):
- United Kingdom (5):
  - Royal Sussex County Hospital, Eastern Road,, Brighton
  - St Marks Hospital, Harrow
  - North Middlesex University Hospital, London
  - St Thomas' Hospital, Lambeth Palace Road, London
  - Stepping Hill Hospital, Stockport